CLINICAL TRIAL: NCT01593137
Title: A Long-term, Randomized, Open-labeled, Parallel-group Trial to Compare the Effects of Liraglutide and Sulphonylurea (Glimepiride) Both in Combination With Metformin on Clinical, Endothelial and Image Markers of Cardiovascular Risk in Patients With Type 2 Diabetes
Brief Title: A Long-term Trial to Compare the Effects of Liraglutide and Sulphonylurea (Glimepiride) Both in Combination With Metformin on Clinical, Endothelial and Image Markers of Cardiovascular Risk in Patients With Type 2 Diabetes
Acronym: ADELANTE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of patients with the criteria established in the protocol.
Sponsor: Fundación Fernández-Cruz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: FFC-0001; 2012-000311-87 (EudraCT Number)
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide; Metformin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide + metformin (Experimental)
  Interventions: Drug: Liraglutide + metformin
- glimepiride + metformin (Active Comparator)
  Interventions: Drug: Glimepiride + metformin

INTERVENTIONS:
Drug: Liraglutide + metformin — Liraglutide 1.8 mg/day + metformin >1500mg/day. Liraglutide will be administered once daily by subcutaneous injection, either in the abdomen, thigh or upper arm.
  Patients will continue on metformin therapy as they were prescribed before enrolment.
  Arms: Liraglutide + metformin
Drug: Glimepiride + metformin — Glimepiride 4 mg/day + metformin >1500 mg/day. Tablets should be swallowed whole with some liquid before or during a substantial breakfast or, if none is taken, shortly before or during the first main meal.
  Patients will continue on metformin therapy as they were prescribed before enrolment.
  Arms: glimepiride + metformin

SUMMARY:
The process of atherosclerosis is multifactorial and involves many mechanisms. The majority of published works have identified endothelial dysfunction as the first step in a cascade of events that culminates in plaque formation. Among the various mechanisms that occur following the attack on the vessel wall, it is thought that stem cells in the form of endothelial progenitor cells (EPCs) are the endothelial protection mechanism.

Factors identified as cardiovascular risk factors, or rather those conditions which suppose a threat to the vessel wall, should therefore be associated with low levels of EPCs. To date this link has been shown in hypertension, diabetes, hyperlipidaemia, and smoking. Furthermore, the lack of wall protection in situations of low levels of EPCs is clearly a biomarker of cardiovascular morbidity and mortality.

On the other hand, the correction of a risk factor allows recuperation of EPCs and is therefore showing itself to be a promising tool for measuring therapeutic efficacy.

The tools for correcting EPC levels are not clearly defined. The effect of statins on levels of EPC has been shown, and the low levels of EPCs in diabetes seem to be susceptible to treatment with statins.

The role of glucagon-like peptide (GLP-1) is slowly being elucidated but the actual mechanism of its potential endothelial protection is unknown, and its effect on EPCs has not been studied.

Liraglutide, a long-acting GLP-1 analogue, could also be an interesting option for long-term vessel wall protection, but to date its ability to correct cardiovascular biomarkers such as EPCs has not been studied.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent obtained before any trial-related activities (trial-related activities are any procedures that would not have been performed during normal management of the subject).
* Male or female patients between 18 and 75 years old;
* Subjects diagnosed with type 2 diabetes for more than 1 year
* Insulin naïve subjects (Allowed are: Previous short term insulin treatment < 28 days in total; Treatment during hospitalisation or during gestational diabetes is allowed for periods < 14 days in total)
* Subjects previously treated with metformin at a minimum dose of 1500 mg/day
* HbA1c from 7% to 9%
* Adherence to injection therapy

Exclusion Criteria:

* Type 1 diabetic patients;
* Use of a GLP-1 receptor agonist (exenatide, liraglutide or other), pramlintide, thiazolidinediones or any DPP-4 inhibitor within the 3 months prior to screening;
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (or their partners). Adequate contraceptive measures are considered the use of hormonal based contraceptives in combination with a barrier contraception,
* Patients with a clinical history of serious cardiovascular events in the last 3 months (myocardial infarction, unstable angina, cerebral infarction, TIA, peripheral arteriopathic event);
* Suspected or confirmed acute pancreatitis;
* Personal history of medullary thyroid carcinoma;
* Patients with congestive heart failure (NYHA I-IV);
* Moderate or severe renal failure (creatinine clearance < 60 ml/min);
* Patients with hepatic failure. This is AST or ALT > 3 times the upper limit of normal, history of cirrhosis or hepatitis;
* Patients with cancer in the last 10 years;
* Patients with terminal diseases;
* Patients unlikely to comply with trial procedures;
* Known psychiatric disease which may interfere with study procedure;
* Any other pathology which may interfere with the study results at the investigator's discretion;
* Known or suspected contraindications to or history of hypersensitivity to the trial product or related products;
* Previous participation in this trial i.e. randomised;
* The receipt of any investigational product within 30 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
assess the effect of treatment with liraglutide compared to glimepiride, as add-on to metformin, for one year on circulating levels of EPCs in patients with type 2 diabetes poorly controlled. | 1 year

SECONDARY OUTCOMES:
assess the efficacy of liraglutide compared to glimepiride, as add-on to metformin, with regards to other surrogate biomarkers of cardiovascular risk: IMT, Central BP, CD40L, hsCRP, Lp-PLA2, BNP. | 1 year
Relationship between EPC levels and all these biomarkers in patients treated with liraglutide compared to those treated with glimepiride. | 1 year
Safety parameters of glycaemic control: HbA1c, FPG | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Calle, MD, Principal Investigator — Hospital Clínico San Carlos, Department of Endocrinology, Metabolism and Nutrition, Spain
Locations (1):
- Hospital Clínico San Carlos, Madrid, Madrid, Spain